CLINICAL TRIAL: NCT04801277
Title: Efficacy of PC6 Electroacupuncture in the Prevention of Nausea Vomiting in Caesarean Patient Under Spinal Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Chan See Yun, Obstetric Anaesthesiologist and acupuncturist, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-19-3279-51524
Record Dates: First submitted 2020-12-07; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Electroacupuncture; Nausea vomiting; Caesarean Delivery
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Randomized double blinded
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture on PC6 and LI4 (Active Comparator): Acupuncture on bilateral acupoints, that are PC6 and LI4. The pericardium meridian PC6 point (Neiguan) is defined as follows. The patient's four fingerbreadths will be placed on the medial aspect of their forearm with the edge of the 4th finger on the wrist crease. This is then subtracted from the width of the interphalangeal joint of her thumb. The point between the tendons of extensor carpi radialis and palmaris longus was the pericardium meridian PC6 point (Neiguan). The large intestine LI4 point (Hegu) located on the dorsum of the hand, between the first and second metacarpal bones, at the midpoint of the second metacarpal bone and close to its radial border.
  Interventions: Procedure: Electroacupuncture on acupoints vs sham points
- Acupuncture on Sham acupoints (Sham Comparator): Acupuncture on bilateral non acupoints. In sham/placebo group, patient will have the acupuncture needles inserted at non-acupoint 2cm radial to PC6 and between 2nd and 3rd metacarpal bone bilaterally, superficial skin piercing (adequate depth to let patient feels needle is inserted)
  Interventions: Procedure: Electroacupuncture on acupoints vs sham points

INTERVENTIONS:
Procedure: Electroacupuncture on acupoints vs sham points — Randomized double blinded clinical trial

SUMMARY:
To determine the ability of electroacupuncture on PC6 versus sham acupuncture in reducing incidence of intraoperative and postoperative nausea vomiting in parturients who underwent Caesarean delivery under spinal anaesthesia

DETAILED DESCRIPTION:
Caesarean rate in most countries are increasing year by year. A report shows that the caesarean section rate for government hospitals in Malaysia was 10.5% in 2000 and 11.0% in 20011 and it rises to 25% of total delivery in Hospital Raja Permaisuri Bainun, Malaysia in year 2018. Nowadays, about 7% of all surgical procedures worldwide are caesarean section and the majority of them are performed with neuraxial blockade, ie epidural anesthesia, spinal anesthesia, or a combined spinal-epidural anesthesia (CSE).

Nausea and vomiting are common intraoperative and postoperative complications in women having caesarean section under neuraxial anesthesia.Compared to the plethora of literatures about PONV, little attention has been paid to nausea vomiting occurring during or after regional anesthesia. These techniques gain increasing attention.

Current literature review indicates a high incidence of IONV during CS under spinal anesthesia up to 80%4. The etiology of intraoperative and postoperative nausea and vomiting (IONV and PONV) is multifactorial. Pregnant women are already likely to suffer from nausea and vomiting because of the pregnancy itself. According to Apfel's score predictive of PONV score that consists of four ascertained risk factors (female, non-smoker, opioid use, previous PONV events or motion sickness), parturients often meet at least two of these criteria with their gender and non-smoker status.

Despite the practice of prescribing antiemetic prophylaxis medication, the incidence of nausea and vomiting in CS patient is still up to 30-50%6. The efficacy of antiemetic drugs is limited and their administration is not free from side effects. Nausea and vomiting not only causes dehydration, electrolyte imbalance and adversely affects wound healing, but also leads to increased wound pain, discomfort, and anxiety among post partum patient. This may further lead to increased medical expenses and extended hospital stay, leaving patient with the overall negative surgical experience. Hence, the idea of multimodal therapy in prophylaxis of IONV and PONV arises.

Non-pharmacological techiniques such as acupuncture, acupressure,and transcutaneous acupoint electrical stimulation of the pericardium 6(PC6) Neiguan point have been studied for the prevention of PONV. The increasing popularity of these modalities is, in part, due to their low cost, simplicity, and in obstetrics, concern about placental transfer and secretion in breast milk of drugs.

It is hypothesized that PC6 electroacupunture stimulation will reduce the incidence of IONV and PONV and reduce the usage of antiemetic drugs in post partum patient.

ELIGIBILITY:
Inclusion Criteria:

* Parturients (36-42 weeks pregnant) aged 18-45 undergoing planned for Caesarean Section.
* American Society of Anaesthesiology class II patients only

Exclusion Criteria:

* Patients with a previous history of PONV or nausea and vomiting in the preceding 24 hours
* Patients who required emergent surgery where delay is inappropriate and can compromise mother and foetus, e.g. foetal distress, foetal bradycardia, chorioamnionitis, cord prolapse, severe preeclampsia
* Patients with documented or known history of allergy to granisetron
* Morbid obesity (BMI>40) as morbid obesity patient will be not be given intrathecal morphine due to increase risk of post operative respiratory depression.
* Patients using any antiemetic drug including dexamethasone for 24 hours prior to Caesarean section (CS)
* Patient who had an implanted pacemaker or defibrillator device. (safety of the use of electroacupuncture on these patient is questionable)
* Patient who received opioids prior to CS (opioid is known to have nausea and vomiting side effect)
* Patient refusal
* Severe preeclampsia, gestational diabetes mellitus on treatment, neurological or cardiac disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative nausea vomiting | Intraoperative 2 hours
  Change in incidence
Postoperative nausea vomiting | Immediate post operative
  Change in incidence
Postoperative nausea vomiting | 12 hours post operative
  Change in incidence
Postoperative nausea vomiting | 24 hours post operative
  Change in incidence

CONTACTS AND LOCATIONS:
Overall Officials: See Yun Chan, Principal Investigator — Hospital Raja Permaisuri Bainun Ipoh
Locations (1):
- Hospital Raja Permaisuri Bainun Ipoh, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No
Study Methodology

REFERENCES:
- [Background] Macario A, Weinger M, Truong P, Lee M. Which clinical anesthesia outcomes are both common and important to avoid? The perspective of a panel of expert anesthesiologists. Anesth Analg. 1999 May;88(5):1085-91. doi: 10.1097/00000539-199905000-00023. PMID 10320175
- [Background] Jelting Y, Klein C, Harlander T, Eberhart L, Roewer N, Kranke P. Preventing nausea and vomiting in women undergoing regional anesthesia for cesarean section: challenges and solutions. Local Reg Anesth. 2017 Aug 9;10:83-90. doi: 10.2147/LRA.S111459. eCollection 2017. PMID 28860857
- [Result] Balki M, Carvalho JC. Intraoperative nausea and vomiting during cesarean section under regional anesthesia. Int J Obstet Anesth. 2005 Jul;14(3):230-41. doi: 10.1016/j.ijoa.2004.12.004. PMID 15935649
- [Result] Arnberger M, Stadelmann K, Alischer P, Ponert R, Melber A, Greif R. Monitoring of neuromuscular blockade at the P6 acupuncture point reduces the incidence of postoperative nausea and vomiting. Anesthesiology. 2007 Dec;107(6):903-8. doi: 10.1097/01.anes.0000290617.98058.d9. PMID 18043058
- [Result] Pierre S, Benais H, Pouymayou J. Apfel's simplified score may favourably predict the risk of postoperative nausea and vomiting. Can J Anaesth. 2002 Mar;49(3):237-42. doi: 10.1007/BF03020521. PMID 11861340

DOCUMENTS (2):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT04801277/Prot_000.pdf
  • Informed Consent Form (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT04801277/ICF_001.pdf